CLINICAL TRIAL: NCT04842175
Title: Evaluation of Education and Equipment of Paramedics in the Prehospital Setting. A Online Based Survey. The EVAIR-Study
Brief Title: Evaluation of Education and Equipment in the Prehospital Setting
Acronym: EVAIR
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, PD Dr. med. Marc Kriege, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUT
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Airway Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a national online based survey the investigators are targeting paramedics for these survey that are involved in prehospital setting. In this study the investigators want to get more information about the current standard or levels of education in prehospital emergency medicine (e.g. airway management) and the incidence of the independently application in daily practice. Furthermore the investigators want to know the current hygiene concepts especially in the actual SARS-CoV-2 Pandemic.

DETAILED DESCRIPTION:
Every participant can answer the survey just once.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants/paramedics

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthy paramedics in Germany
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Perception of intubation success | through study completion, on average 1 Month
  incidence of failed intubation attempts

SECONDARY OUTCOMES:
Perception of hygiene concepts in SARS-CoV-2 Pandemic | through study completion, on average 1 Month
  face masks, gloves face shields for hygiene concept

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, PhD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany